CLINICAL TRIAL: NCT06988137
Title: Comparative Evaluation of Kinesio Taping, Buddy Taping, and Splinting in Finger Injuries: A Randomized Controlled Trial
Brief Title: Kinesio Taping for Finger Injuries
Acronym: KT Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onur Gültekin (Other)
Responsible Party: Sponsor-Investigator, Onur Gültekin, Orthopaedic Surgeon, Fatih Sultan Mehmet Training and Research Hospital
Organization: Fatih Sultan Mehmet Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSMEAH-2022-78-KT
Record Dates: First submitted 2025-05-14; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Finger Fracture; Finger Sprain; Ligament Injury of the Finger; Proximal Interphalangeal (PIP) Joint Injury
Keywords: Kinesio taping; Buddy taping; Conservative treatment; QuickDASH; Grip strength; Range of motion; Non-operative hand fracture; Randomized controlled trial
MeSH Terms: interventions — Splints

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three treatment groups (Kinesio taping, buddy taping, or splinting) and followed for 3 months.
Who Masked: Outcomes Assessor
Masking Description: Outcomes were assessed by an independent orthopedic surgeon blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Taping Group (Experimental): Participants received Kinesio taping using the ligament correction technique with 75-100% elasticity. Immediate active motion was encouraged without immobilization.
  Interventions: Device: Kinesio Taping
- Buddy Taping (Active Comparator): Participants received buddy taping with adjacent finger stabilization and interdigital padding. Mobilization was allowed after 2 weeks.
  Interventions: Procedure: Buddy Taping
- Splinting Group (Active Comparator): Participants were treated with a static volar splint immobilizing the PIP and DIP joints at 20° flexion.
  Interventions: Device: Splinting

INTERVENTIONS:
Device: Kinesio Taping — Elastic therapeutic tape was applied using the ligament correction technique. The tape was reapplied at Day 3 and Day 21 under supervision
  Arms: Kinesio Taping Group
Procedure: Buddy Taping — Buddy taping involved strapping the injured finger to an adjacent digit using medical tape. Early motion was restricted.
  Arms: Buddy Taping
Device: Splinting — A custom-molded thermoplastic splint was applied to restrict joint movement and maintain alignment. Patients remained immobilized until Week 3.
  Arms: Splinting Group

SUMMARY:
This study is a prospective, randomized controlled trial evaluating the effectiveness of three conservative treatment approaches-Kinesio taping (KT), buddy taping (BT), and static splinting-for managing finger ligament injuries and non-displaced fractures. A total of 175 patients between the ages of 5 and 60 were randomly assigned to one of the treatment groups and monitored over a 3-month period. The study aims to assess outcomes including range of motion (ROM), grip strength, pain levels, and functional recovery using the QuickDASH questionnaire.

DETAILED DESCRIPTION:
Finger ligament injuries and non-displaced fractures are common conditions encountered in both pediatric and adult orthopedic populations. Conservative treatment options such as buddy taping and splinting are commonly employed in clinical practice, although each method may affect mobility and patient comfort differently.

This randomized controlled trial was conducted to evaluate three conservative treatment modalities-Kinesio taping (KT), buddy taping (BT), and static volar splinting-in patients aged 5 to 60 years. Participants were randomly assigned to one of the three treatment groups and evaluated at three time points: Day 3, Week 3, and Month 3.

The primary outcome measure was the range of motion of the injured finger. Secondary outcomes included grip strength, pain scores, QuickDASH assessments, and incidence of skin-related complications. Outcome evaluations were performed by an independent orthopedic surgeon who was blinded to group assignment.

Patients were stratified into pediatric and adult subgroups to assess age-related differences in treatment response. The study followed a parallel assignment design and employed single-blind outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 60 years
* Presentation within 5 days of injury
* Acute finger ligament sprain or non-displaced finger fracture (PIP or phalangeal)
* Ability to provide informed consent (or parental consent for minors)
* Availability for 3-month follow-up

Exclusion Criteria:

* Open fractures
* Polytrauma or systemic injury
* Delayed presentation (>5 days post-injury)
* Need for surgical fixation
* Previous injury or deformity in the same finger
* Neurological or rheumatologic disorders affecting hand function

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Range of Motion (ROM) in Injured Finger | Week 3 and Month 3
  Flexion and extension angles of the injured finger joints measured using a digital goniometer. Results expressed in degrees. Higher values indicate better mobility.

SECONDARY OUTCOMES:
QuickDASH Disability Score | Week 3 and Month 3
  Functional status of the upper limb evaluated using the QuickDASH questionnaire. Scores range from 0 (no disability) to 100 (maximum disability). Lower scores indicate better function.
Grip Strength Recovery | Month 3
  Hand grip strength of the injured side measured using a dynamometer, expressed as a percentage of the unaffected side. Higher percentages indicate better recovery.
Incidence of Skin Complications | Up to Month 3
  Occurrence of skin maceration, irritation, or pressure sores recorded during follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations, lack of specific participant consent for data sharing beyond the study scope, and the absence of a secure data repository. The study was conducted at a single institution and was not originally designed for secondary data use. Future data sharing may be considered upon formal request and appropriate ethical approvals.